CLINICAL TRIAL: NCT03556865
Title: Knowledge, Attitude, And Practice In A Group Of Egyptian Dentists Towards Preventive Measures In Pediatric Dentistry: A Cross-Sectional Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, MANAR SAID ABDEL HAFIZ AL SHARIF, Manar Al Sharif, Cairo University
Other Study IDs: MSHARIF
Record Dates: First submitted 2018-06-04; First posted 2018-06-14 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: A self administered questionnaire — The questionnaire is in English language, it contains binary questions related to KAP on different preventive measures in pediatric dentistry and consists of 38 items divided into 4 sections as follows:
  I) Socio-demographic data: (7 items). It includes gender, total years in practice, nature of primary practice, school of graduation, scientific degree and specialty II) Assessment of Knowledge towards preventive measures in pediatric dentistry. (16 items) III) Assessment of Attitude towards preventive measures in pediatric dentistry. (10 items) IV) Assessment of Practice towards preventive measures in pediatric dentistry. (5items) One score is given for each response to items.

SUMMARY:
The study will include general dental practitioners or dental specialists from Police Academy Hospital and pediatric dentists from Pediatric dentistry department at Faculty of Dentistry Cairo University.

A self-administered questionnaire will be given to dentists by direct interviewing and they will be allowed to complete the questionnaire in Faculty of Dentistry, Cairo University or Police Academy Hospital. The data will be based on a collection of responses to the 38 items in the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Egyptian dentists working in either Faculty of Dentistry Cairo University or Police Academy Hospital.
* Postgraduate students.

Exclusion Criteria:

* Refusal to participate in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Egyptian dentists working in either Faculty of Dentistry Cairo University or Police Academy Hospital and postgraduate students at Faculty if Dentistry - Cairo University
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Knowledge,attitude and practice towards preventive measures in pediatric dentistry. | 3 months
  Measuring device is a KAP questionnaire and measuring unit id binary questions

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol